CLINICAL TRIAL: NCT02811159
Title: An Open-Label Extension Study of 12 mg Proellex® (Telapristone Acetate) Administered Orally in the Treatment of Premenopausal Women With Confirmed Symptomatic Uterine Fibroids
Brief Title: An Extension Study of 12 mg Proellex® (Telapristone Acetate) Administered Orally in the Treatment of Premenopausal Women With Confirmed Symptomatic Uterine Fibroids
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZPU-203EXT
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma | interventions — telapristone acetate

ARMS (1):
- Telapristone Acetate 12 mg (Experimental): Telapristone acetate 12 milligrams (mg), orally, once daily for two 18-weeks courses (Treatment Courses 1 and 2) separated by an off-drug interval (ODI).
  Interventions: Drug: Telapristone acetate

INTERVENTIONS:
Drug: Telapristone acetate — Telapristone acetate, orally, once daily for three 18-weeks courses separated by an ODI.
  Other Names: Proellex®

SUMMARY:
To determine the safety of extended treatment with Proellex® in women who have successfully completed either study ZPV-201 [NCT02323646] or ZPU-203 [NCT02301897] and meet eligibility criteria.

DETAILED DESCRIPTION:
This study will be for participants who had completed either ZPV-201 or ZPU-203.

ELIGIBILITY:
Inclusion Criteria:

* Completed either study ZPV-201 [NCT02323646] or ZPU-203 [NCT02301897]
* Agreement not to attempt to become pregnant during the trial
* Agreement to use alcohol in moderation and record the daily consumption (note: elevated liver enzymes may result in discontinuation from the study)
* Ability to complete a daily subject diary and study procedures in compliance with the protocol
* Women of child-bearing potential must be willing to use double-barrier contraception during the study and off-drug intervals. Acceptable double-barrier methods are: male condom with spermicide; male condom with diaphragm; diaphragm containing spermicide plus additional intra-vaginal spermicide
* Has a negative pregnancy test at Visit 1
* Subject is available for all treatment and follow-up visits

Exclusion Criteria:

* Subject had a significant decrease in bone mineral density while participating in ZPV-201 or ZPU-203 (total hip or spine measurement decreased by 5% or more)
* Subject has undergone hysterectomy and/or bilateral oophorectomy since enrollment in ZPV-201 or ZPU-203
* Subject is pregnant or lactating or is attempting or expecting to become pregnant during the entire study period
* Subjects with abnormally high liver enzymes or liver disease. [alanine aminotransferase (ALT) or aspartate aminotransferase (AST) exceeding 2 x upper limit of normal (ULN) and total bilirubin exceeding 1.5 x ULN at Visit 1 and confirmed on repeat].
* Subject has a hemoglobin of <7.5 grams per deciliter (g/dL) at Visit 1
* Concurrent use of any testosterone, progestin, androgen, estrogen, anabolic steroids, dehydroepiandrosterone (DHEA) or hormonal products for at least 2 weeks prior to Visit 1
* Use of oral contraceptives in the 30 days preceding screening. Use of Depo-Provera® in the preceding 10 months
* Use of Gonadotrophin releasing hormone agonist (GnRHas) (e.g. Lupron Depot) within 3 months prior to screening (Lupron Depot must have a wash-out period of 3 months prior to screening)
* Has an intra-uterine device (IUD) in place
* Current cervical dysplasia classified as Atypical Squamous Cells of Undetermined Significance (ASCUS) associated with high-risk human papilloma virus (HPV)
* Current diagnosis of Low/High Grade Squamous Intraepithelial Lesion (LGSIL or HGSIL), endometrial polyps or hyperplasia
* Observation or history of abnormal endometrial biopsy including the presence of endometrial intraepithelial neoplasia (EIN)
* Recent history (within past 6 months) of alcoholism or drug abuse
* Endometrial stripe ≥18 mm in thickness at Visit 1 (subject may be enrolled with sponsor approval)
* Subject is currently taking cimetidine or spironolactone or has taken them in the last 30 days
* Clinically significant abnormal findings on Visit 1 examination and laboratory assessments or any condition which in the opinion of the investigator would interfere with the subject's ability to comply with the study instructions or endanger the subject if she took part in the study.

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07-26 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chan, Study Director — Allergan
Locations (8):
- United States (8):
  - KO Clinical Research, LLC, Fort Lauderdale, Florida
  - Atlanta Women's Research Institute, Inc., Atlanta, Georgia
  - WR-Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - Southern Clinical Research Associates, LLC, Metairie, Louisiana
  - The Jackson Clinic, PA, Jackson, Tennessee
  - Advances in Health, Houston, Texas
  - The Women's Hospital of Texas Clinical Research Center, Houston, Texas
  - Clinical Research Partners, LLC, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who had successfully completed either study ZPV-201 [NCT02323646] or ZPU-203 [NCT02301897] were enrolled in this study.
Groups:
- Telapristone Acetate 12 mg: Telapristone acetate 12 mg, orally, once daily for two 18-weeks courses (Treatment Courses 1 and 2) separated by an off-drug interval (ODI).
Period: Treatment Course 1
Arm/Group | Telapristone Acetate 12 mg
Started | 20
Completed | 19
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: Treatment Course 2
Arm/Group | Telapristone Acetate 12 mg
Started | 4 (Not all participants who completed the Treatment Course 1 entered the Treatment Course 2.)
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all study participants who were randomized, received study drug and had some post-baseline safety data.
Arm/Group | Telapristone Acetate 12 mg
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Safety population included all study participants who were randomized, received study drug and had some post-baseline safety data.
  years | 43.3 (3.62)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Safety population included all study participants who were randomized, received study drug and had some post-baseline safety data.
  Participants
    Female | 20
    Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Amenorrhea
Description: Amenorrhea was defined as no bleeding intensity score greater than 1 using the Daily Diary Card during the 28 days leading up to the last day of dosing at Week 18. Bleeding intensity was graded on a 5-point scale where: 0=no bleeding to 4=heavy bleeding.
Time Frame: At the end of 18 weeks Treatment Course 1
Population: Intent-to-treat (ITT) population included all participants who received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Telapristone Acetate 12 mg
Number analyzed (Participants) | 20
percentage of participants | 35.00
Statistical Analysis 1: Comparison: Telapristone Acetate 12 mg; Test type: Other; p = 0.1797, Chi-Square Test

2. Primary Outcome: Percentage Change From Baseline in Total Uterine Fibroid System Quality of Life Survey System Severity (UFS-SSS) Score
Description: UFS-SSS is an 8-question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. Each question was answered on a 5-point scale where 1=Not at all to 5=A very great deal. The sum of the total scores was transformed to a range of 0=no symptoms (best) to 100=most severe symptoms (worst). A negative percentage change from Baseline indicates improvement.
Time Frame: Baseline to the end of 18-weeks Treatment Course 1
Population: ITT population included all participants who received study drug.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Telapristone Acetate 12 mg
Number analyzed (Participants) | 20
percent change | -7.21 (20.046)
Statistical Analysis 1: Comparison: Telapristone Acetate 12 mg; Test type: Other; p = 0.1250, Wilcoxon Signed-Rank Test

3. Primary Outcome: Percentage Change From Baseline in the Individual UFS-SSS Subscale Score Question 1
Description: UFS-SSS is an 8-question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 1: During the previous 3 months how distressed were you by "heavy bleeding during your menstrual period"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: Baseline to the end of 18-weeks Treatment Course 1
Population: ITT population included all participants who received study drug.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Telapristone Acetate 12 mg
Number analyzed (Participants) | 20
percent change | -10.50 (26.253)
Statistical Analysis 1: Comparison: Telapristone Acetate 12 mg; Test type: Other; p = 0.2500, Wilcoxon Signed-Rank Test

4. Primary Outcome: Percentage Change From Baseline in the Individual UFS-SSS Subscale Score Question 2
Description: UFS-SSS is an 8-question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 2: During the previous 3 months how distressed were you by "passing blood clots during your menstrual period"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: Baseline to the end of 18-weeks Treatment Course 1
Population: ITT population included all participants who received study drug.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Telapristone Acetate 12 mg
Number analyzed (Participants) | 20
percent change | -5.83 (18.157)
Statistical Analysis 1: Comparison: Telapristone Acetate 12 mg; Test type: Other; p = 0.5000, Wilcoxon Signed-Rank Test

5. Primary Outcome: Percentage Change From Baseline in the Individual UFS-SSS Subscale Score Question 3
Description: UFS-SSS is an 8-question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 3: During the previous 3 months how distressed were you by "fluctuation in the duration of your menstrual period compared to your previous cycle"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: Baseline to the end of 18-weeks Treatment Course 1
Population: ITT population included all participants who received study drug.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Telapristone Acetate 12 mg
Number analyzed (Participants) | 20
percent change | -8.75 (23.333)
Statistical Analysis 1: Comparison: Telapristone Acetate 12 mg; Test type: Other; p = 0.2500, Wilcoxon Signed-Rank Test

6. Primary Outcome: Percentage Change From Baseline in the Individual UFS-SSS Subscale Score Question 4
Description: UFS-SSS is an 8-question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 4: During the previous 3 months how distressed were you by "fluctuation in the length of your monthly cycle compared to your previous cycles"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: Baseline to the end of 18-weeks Treatment Course 1
Population: ITT population included all participants who received study drug.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Telapristone Acetate 12 mg
Number analyzed (Participants) | 20
percent change | -3.75 (16.771)
Statistical Analysis 1: Comparison: Telapristone Acetate 12 mg; Test type: Other; p = 1.0000, Wilcoxon Signed-Rank Test

7. Primary Outcome: Percentage Change From Baseline in the Individual UFS-SSS Subscale Score Question 5
Description: UFS-SSS is an 8-question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 5: During the previous 3 months how distressed were you by "feeling tightness or pressure in your pelvic area"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: Baseline to the end of 18-weeks Treatment Course 1
Population: ITT population included all participants who received study drug.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Telapristone Acetate 12 mg
Number analyzed (Participants) | 20
percent change | -4.17 (33.278)
Statistical Analysis 1: Comparison: Telapristone Acetate 12 mg; Test type: Other; p = 0.8750, Wilcoxon Signed-Rank Test

8. Primary Outcome: Percentage Change From Baseline in the Individual UFS-SSS Subscale Score Question 6
Description: UFS-SSS is an 8-question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 6: During the previous 3 months how distressed were you by "frequent urination during the daytime hours"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: Baseline to the end of 18-weeks Treatment Course 1
Population: ITT population included all participants who received study drug.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Telapristone Acetate 12 mg
Number analyzed (Participants) | 20
percent change | -7.33 (22.675)
Statistical Analysis 1: Comparison: Telapristone Acetate 12 mg; Test type: Other; p = 0.5000, Wilcoxon Signed-Rank Test

9. Primary Outcome: Percentage Change From Baseline in the Individual UFS-SSS Subscale Score Question 7
Description: UFS-SSS is an 8-question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 7: During the previous 3 months how distressed were you by "frequent night time urination"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: Baseline to the end of 18-weeks Treatment Course 1
Population: ITT population included all participants who received study drug.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Telapristone Acetate 12 mg
Number analyzed (Participants) | 20
percent change | 6.67 (35.210)
Statistical Analysis 1: Comparison: Telapristone Acetate 12 mg; Test type: Other; p = 0.5000, Wilcoxon Signed-Rank Test

10. Primary Outcome: Percentage Change From Baseline in the Individual UFS-SSS Subscale Score Question 8
Description: UFS-SSS is an 8-question assessment tool used to measure symptom severity and has been validated as a three month look back questionnaire. The participant answered UFS-SSS subscale question 8: During the previous 3 months how distressed were you by "feeling fatigued"? using a 5-point scale where 1=Not at all to 5=A very great deal. A negative percentage change from Baseline indicates improvement.
Time Frame: Baseline to the end of 18-weeks Treatment Course 1
Population: ITT population included all participants who received study drug.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Telapristone Acetate 12 mg
Number analyzed (Participants) | 20
percent change | -6.67 (16.579)
Statistical Analysis 1: Comparison: Telapristone Acetate 12 mg; Test type: Other; p = 0.2500, Wilcoxon Signed-Rank Test

11. Primary Outcome: Change From Baseline in Pictorial Blood Loss Assessment Chart (PBAC) Score
Description: Uterine bleeding was assessed with the use of the PBAC, a validated self-reporting method to estimate menstrual blood loss. Participants recorded daily the number of tampons and towels used and the degree to which individual items were soiled with blood (plus small or large clots). Pictorial scores range from score 1 for slightly stained tampon/towel, 5 for a partially stained tampon/towel, 10 for a completely saturated tampon, 20 for a completely saturated towel, and 5 for each episode of flooding and for each blood clot larger than a quarter in size. Total score can range from 0 (no bleeding) to >500. Higher scores indicate more bleeding. Lower scores indicate less bleeding. A negative change from Baseline indicates improvement (reduction in bleeding).
Time Frame: Baseline to the end of 18-weeks Treatment Course 1
Population: ITT population Included all participants who received study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telapristone Acetate 12 mg
Number analyzed (Participants) | 20
score on a scale
  Baseline | 139.50 (196.111)
  Change from Baseline to Week 18 Course 1 | -81.10 (239.790)
Statistical Analysis 1: Comparison: Telapristone Acetate 12 mg; Test type: Other; p = 0.0645, Wilcoxon Signed-Rank Test

12. Primary Outcome: Percentage Change From Baseline in Total Uterine Fibroid Volume
Description: The total uterine fibroid volume was measured by Magnetic Resonance Imaging (MRI). A negative percentage change from Baseline indicates improvement.
Time Frame: Baseline to the end of 18-weeks Treatment Course 1
Population: ITT population Included all participants who received study drug. MRI data was only available for 3 participants.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Telapristone Acetate 12 mg
Number analyzed (Participants) | 3
percent change | 0.00 (0.000)

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 30 days after the last dose of study drug (approximately 43 weeks)
Description: Safety population consisted of all study participants who were randomized, received study drug and had some post-baseline safety data.
Arm/Group | Telapristone Acetate 12 mg
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 11/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telapristone Acetate 12 mg (N=20)
Liver function test abnormal (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telapristone Acetate 12 mg (N=20)
Abdominal pain (Gastrointestinal disorders) | 1
Diverticulitis (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Hot flush (General disorders) | 2
Chills (General disorders) | 1
Fatigue (General disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Acute sinusitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1
Blood cholesterol increased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Disorientation (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Endometrial hypertrophy (Reproductive system and breast disorders) | 2
Menometrorrhagia (Reproductive system and breast disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT02811159/Prot_SAP_000.pdf